CLINICAL TRIAL: NCT04854772
Title: Mind Body Intervention for COVID-19 Long Haul Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Michael Donnino, Professor of Emergency Medicine, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021P-000336
Record Dates: First submitted 2021-04-20; First posted 2021-04-22 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: COVID-19 Long Haul Syndrome

STUDY DESIGN:
Intervention Model Description: Feasibility/pilot Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mind Body Syndrome Therapy for Long Covid (Experimental): The participants will receive an initial one-on-one interview, followed by 1 to 2 hour biweekly group interactive, educational sessions for 12 weeks. This program also includes a day-long "retreat" at the end of the required course period. Participants will also be provided reading materials to study during the intervention period
  Interventions: Behavioral: Mind Body Syndrome Therapy for Long Covid

INTERVENTIONS:
Behavioral: Mind Body Syndrome Therapy for Long Covid — The intervention consists of a mind-body based intervention for the COVID long haul syndrome. The components of the intervention include knowledge therapy, desensitization, emotional expression, and stress reduction techniques.

SUMMARY:
The present study is a feasibility study in which we will determine if a mind-body program that we have previously developed for chronic back pain can improve the multiple somatic complaints associated with the COVID Long Haul Syndrome.

DETAILED DESCRIPTION:
This study is a pilot and feasibility study to determine if a mind-body program that we have previously developed for chronic back pain can improve the multiple somatic complaints associated with the COVID Long Haul Syndrome in patients without evidence of ongoing tissue injury. We will perform a 12-week intervention consisting of a series of classes which will focus on knowledge therapy, desensitization, emotional expression, and stress reduction.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient ≥ 18 years old
* New symptoms attributed to the post-covid long-haul syndrome (extremity pain, dyspnea, headaches, chest pain, fatigue) occurring after an acute phase of COVID19
* Minimum of at least 12 weeks after the end of the acute phase of COVID-19 infection
* Persistence of symptoms for a least 1 month with no identified other organic etiology
* Score ≥ 3 or more on the SSS-8 score
* Symptoms present for a minimum of 4 days a week
* Willingness to consider mind-body intervention

Exclusion Criteria:

* Patients < 18 years of age
* Patients > 60 years of age
* Diagnosed (non-COVID-19) organic disease as cause of pain, such as (but not limited) to malignancy, neurologic disorder (i.e., amyotrophic lateral sclerosis), cauda equina syndrome (note that pain related to disc disease is not an exclusion unless there are neurological impairments).
* Patients with previous severe COVID-19 disease, defined as those who had been admitted to the ICU or have objective evidence of ongoing organ injury (e.g., persistent chest radiographic abnormalities or myocarditis)
* Identified lung or cardiac injury in subjects with chest pain or dyspnea (e.g., chest radiograph abnormalities, cardiac ultrasound showing myocarditis or depressed ejection fraction )
* Patients with a diagnosis of significant psychiatric comorbidities such as schizophrenia or dementia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2022-08-09 (Actual)

PRIMARY OUTCOMES:
Change in somatic symptom severity | Baseline, 4, 8, and 13 weeks
  Will be assessed using the Somatic Symptom Scale-8 (SSS-8). The minimum score is 0 and the maximum 32, with higher values indicating a worse outcome (more severe symptoms)

SECONDARY OUTCOMES:
Average Pain | Baseline, 4, 8, and 13 weeks
  Will be assessed using the Brief Pain Inventory (BPI). The minimum score is 0 and the maximum is 10, with higher values indicating higher pain.
Pain intensity | Baseline 4, 8, and 13 weeks
  Will be assessed using the Brief Pain Inventory (BPI). The minimum score is 0 and the maximum is 10, with higher values indicating higher pain.
Pain-related Anxiety | Baseline 4, 8, 13 weeks
  Will be assessed using the Pain Anxiety Symptom Scale (PASS). The minimum score is 0 and the maximum 100, with higher values indicating higher pain anxiety
Fatigue | Baseline 4, 8, 13 weeks
  Will be assessed using the Fatigue Severity Scale (FSS). The minimum score is 9 and the maximum 63, with higher scores indicating greater fatigue severity
Dyspnea | Baseline 4, 8, and 13 weeks
  Will be assessed using the Multidimensional Dyspnea Profile (MDP). A1, Scale: Scale about breathing sensations with a defined start- and endpoint (neutral - unbearable). Values reach from 0-10, and higher values represent a worse outcome.
  SQ1 (sensoric quality), Choice: 5 Phrases and terms about breathing sensations. Choose between yes and no and select one as "most accurately".
  SQ2 (sensoric quality), Scales: 5 subscales about intensity of breathing sensations. Values reach from 0 - 10, and higher values represent a worse outcome.
  A2 (emotional quality), Scales: 5 subscales about emotions. Values reach from 0 - 10, and higher values represent a worse outcome.
Brain Fog | Baseline, 4, 8, and 13 weeks
  Will be assessed using a numerical rating scale (0-5). Higher numbers represent more severe of brain fog
Physical Functioning | Baseline, 4, 8, and 13 weeks.
  Will be assessed using the Patient Reported Outcomes Measurement Information System (PROMIS) The minimum score is 0 and maximum is 16. Higher numbers represent less physical functioning capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Donnino, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Donnino M, Howard P, Mehta S, Silverman J, Cabrera MJ, Yamin JB, Balaji L, Berg KM, Heydrick S, Edwards R, Grossestreuer AV. Psychophysiologic Symptom Relief Therapy (PSRT) for Post-acute Sequelae of COVID-19. Mayo Clin Proc Innov Qual Outcomes. 2023 May 19;7(4):337-48. doi: 10.1016/j.mayocpiqo.2023.05.002. Online ahead of print. PMID 37361483